CLINICAL TRIAL: NCT04842318
Title: Rituximab Maintenance Treatment of Newly Diagnosed Follicular Lymphoma After Induction Therapy of Rituximab Combined With Bendamustine (BR) or Cyclophosphamide, Vincristine, Doxorubicin, Prednisone (RCHOP) or Lenalidomide (R2): a Multicenter Clinical Study
Brief Title: Rituximab Maintenance Treatment of Newly Diagnosed Follicular Lymphoma After BR or RCHOP or R2: a Multicenter Clinical Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL-001
Record Dates: First submitted 2021-04-04; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; Rituximab; maintenance treatment
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BR+R (Experimental): Induction Therapy: Rituximab Combined With Bendamustine Maintenance Treatment: Rituximab
  Interventions: Drug: BR for 6 cycles +R for 8 cycles
- RCHOP+R (Experimental): Induction Therapy: Rituximab Combined With Cyclophosphamide, Vincristine, Doxorubicin, Prednisone Maintenance Treatment: Rituximab
  Interventions: Drug: RCHOP for 6 cycles +R for 8 cycles
- R2+R2 (Experimental): Induction Therapy: Lenalidomide Combined With Rituximab Maintenance Treatment: Lenalidomide Combined With Rituximab
  Interventions: Drug: R2 for 6 cycles + R2 maintenance

INTERVENTIONS:
Drug: BR for 6 cycles +R for 8 cycles — The patients will be given Bendamustine (90mg/m2 d1,2, every 28 days for total 6 courses) combined with Rituximab (375mg/m2 d0, every 28 days for total 6 courses) followed by Rituximab (375mg/m2 d1, every 3 months for total 8 courses)
  Arms: BR+R
Drug: RCHOP for 6 cycles +R for 8 cycles — The patients will be given RCHOP (Rituximab 375mg/m2 ivgtt, D0, Cyclophosphamide 750mg/m2, ivgtt D1, doxorubicin 50mg/m2,ivgtt D1, Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5 every 21 days for total 6 courses) followed by Rituximab (375mg/m2 d1, every 3 months for total 8 courses)
  Arms: RCHOP+R
Drug: R2 for 6 cycles + R2 maintenance — The patients will be given Lenalidomide (25mg/d, po, D1-10, every 21 days for total 6 courses) combined with Rituximab (375mg/m2 d0, every 21 days for total 6 courses) followed by Lenalidomide (25mg/d, po, D1-10, every 28 days for total 6 courses) combined with Rituximab (375mg/m2 d1, every 3 months for total 8 courses)
  Arms: R2+R2

SUMMARY:
This multi-center clinical study will evaluate the efficacy of Rituximab maintenance treatment of newly diagnosed follicular lymphoma after induction therapy of BR, RCHOP or R2.

DETAILED DESCRIPTION:
Follicular lymphoma (FL) is a lymphoma of B cells in follicular center. It is a common pathological subtype of lymphoma, and its incidence rate is only next to diffuse large B cell lymphoma (DLBCL). The initial remission rate is high, but the tumor generally recurrent, making it difficult to be completely cured. This study attempts to explore the efficacy and safety of rituximab monotherapy maintenance after BR, RCHOP, R2 regimen induction therapy in the treatment of follicular patients, and to find the best way to maximize survival benefit and reduce treatment toxicity for FL patients. The study can improve the quality of life, prolong the survival and avoid the transformation to invasive lymphoma in patients with follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed CD20 positive follicular lymphoma grade 1, 2, or 3A based on 2016 WHO classification
* Treatment naive
* Age ≥ 18 years
* Indications for treatment confirmed
* Must has measurable lesion in CT or PET-CT prior to treatment
* Considered suitable for RCHOP, BR or R2 regimens
* Informed consented

Exclusion Criteria:

* Transformed follicular lymphoma or 3B follicular lymphoma;
* HBsAg positive and / or HBcAb positive with HBV DNA titer; HCV antibody positive with HCV-RNA; or HIV positive
* Central nervous system or meninges involved
* Any drug contraindication in the treatment plan
* Patients judged by other researchers to be unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
MRD negative rate of bone marrow at 24 weeks | At 24 weeks
  Percentage of participants with negative MRD estimated by q-RT-PCR of bone marrow

SECONDARY OUTCOMES:
Overall response rate | 21 days after 6 cycles of induction therapy (each cycle is 21 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Progression of disease within 24 months | Baseline up to data cut-off (24 months)
  Progression of disease within 24 months was defined as the rate of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Event-free survival | Baseline up to data cut-off (up to approximately 4 years)
  Event-free survival was defined as the time from the date of diagnosis until the date of the first documented day of events.
Time to Progression | Baseline up to data cut-off (up to approximately 4 years)
  Time to Progression was defined as the time from the date of diagnosis until the date of the first documented day of disease progression, using 2014 Lugano criteria, whichever occurred first.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  Duration of response was defined as the time from the date of diagnosis until the date of the first documented day of disease relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Time to Next Anti-lymphoma Treatment | Baseline up to data cut-off (up to approximately 4 years)
  Time to Next Anti-lymphoma Treatment was defined as the time from the date of first treatment until the date patients need to receive next anti-lymphoma treatment on the basis of investigator assessments according to 2014 Lugano criteria
Progression Free Survival | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 30 days after completion of study treatment
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events
MRD negative rate of peripheral blood at 24 weeks | At 24 weeks
  Percentage of participants with negative MRD estimated by q-RT-PCR of peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No